CLINICAL TRIAL: NCT02792920
Title: Multicenter Registry of Very Early and Late Clinical Outcomes to Everolimus-eluting Cobalt-Chromium Stent In Patients With ST Elevation Myocardial Infarction
Acronym: XIENCE STEMI
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hyogo Brain and Heart Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: XIENCE STEMI Registry
Record Dates: First submitted 2016-03-02; First posted 2016-06-08 (Estimated); Last update posted 2016-06-08 (Estimated); Status verified 2016-06

CONDITIONS: ST-elevation Acute Myocardial Infarction; STEMI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

ARMS (1):
- CoCr-EES (Other)
  Interventions: Device: CoCr-EES

INTERVENTIONS:
Device: CoCr-EES

SUMMARY:
To compare early and late clinical outcomes with everolimus-eluting cobalt-chromium stent in patients with ST-elevation acute myocardial infarction, as well as identify the characteristics and efficacy of CoCr-EES.

Also, OCT sub-analysis will be conducted

ELIGIBILITY:
Inclusion Criteria:

1. Patients with STEMI who are able to undergo CoCr-EES implantation.
2. Patients with no history of PCI in the target vessel
3. Patients who are 20 or older at the time of informed consent
4. Patients who provided written informed consent by himself/herself
5. Patients who are judged by their treating physician to be able to undergo PCI with CoCr-EES
6. Patients for whom thrombus aspiration prior to CoCr-EES implantation can be recommended
7. Patients who meet all the following vascular inclusion criteria i.Patients with target lesion in native coronary artery ii.Patients with visual maximum vessel diameter of the target stent site in target lesion
8. Patients were obtained finally revascularization of TIMI 3 by visual observation in the target vessel
9. Patients who are able to treat with CoCr-EES the diameter 2.5mm or more and 3.5mm or less and the length of 8mm or more and 28mm or less.

Exclusion Criteria:

1. Patients participating in the other ongoing registry or clinical study(except post-marketing surveillance of CoCr-EES), or receiving treatment which may impact on endpoints of this study.
2. Patients presenting with cardiogenic shock
3. Patients for whom 12-month and 36-month CAG and clinical follow up is considered difficult (patient's residence should also be taken into account)
4. Patients with responsible lesion in left main trunk
5. Patients with renal insufficiency or with chronic renal failure with serum creatinine level of 2.0mg/dL or higher at visit
6. Patients on hemodialysis
7. Patients with a known history of adverse drug reactions to aspirin, or clopidogrel or prasugrel (This may not apply if safety of ticlopidine is confirmed as an alternative drug.)
8. Patients who are below the age of 20
9. Women who were positive in pregnancy test or wish to become pregnant during study duration
10. Patients who newly developed AMI attributable to the prior stented site
11. Patients with a known history of allergy to drug, polymer, metal, and other materials used in CoCr-EES
12. Patients diagnosed with hepatic insufficiency
13. Patients with target lesion in saphenous vein graft
14. Patients with active malignant tumor

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-04 (Estimated)

PRIMARY OUTCOMES:
Target vessel failure (TVF) | 12 months
  Target vessel failure (TVF) at 12 months after CoCr-EES implantation. TVF consists of defined as cardiac death, target vessel-related recurrent myocardial infarction (MI) or Target Lesion Revascularization (TLR)

SECONDARY OUTCOMES:
MI (QMI and Non-QMI) | 12 months
Any TLR | 12 months and 36 months
Any Target Vessel Revascularization (TVR) | 12 months and 36 months
Death | 12 months and 36 months
MACE (Cardiac death, MI and TLR) | 12 months and 36 months
Definite or Probable stent thrombosis | 12 months and 36 months

CONTACTS AND LOCATIONS:
Locations (2):
- Japan (2):
  - Hyogo Brain and Heart Center, Himeji, Hyogo,
  - Higashi Takarazuka Sato Hospital, Takarazuka, Hyogo